CLINICAL TRIAL: NCT00801294
Title: A Phase II Trial of Weekly Alternating Sequential Administration of BIBF 1120 and BIBW 2992 in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: 1239.2; EudraCT 2006-000893-56
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nintedanib; Afatinib

INTERVENTIONS:
Drug: BIBF 1120 and BIBW 2992

SUMMARY:
The primary objective of this trial is to explore the overall objective best response rate and the rate of non-progression at 16 weeks of sequential, alternating weekly administration of BIBF 1120 and BIBW 2992 in patients with metastatic CRC based on the RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Signed informed consent.
3. Histologically proven colorectal adenocarcinoma
4. History or presence of metastatic colorectal cancer (stage IV)
5. Measurable (>1 cm) or evaluable tumour deposit (according to RECIST criteria)
6. Documented progression or unacceptable toxicity on the last therapy
7. Progression on oxaliplatin-based chemotherapy or unacceptable residual neurotoxicity on oxaliplatin
8. Progression on irinotecan-based chemotherapy or unacceptable toxicity on irinotecan
9. If patients have been previously exposed to Cetuximab or other EGFR inhibitor, they must have shown progression or unacceptable toxicity
10. If patients have been previously exposed to Bevacizumab or other VEGF inhibitor, they must have shown progression or unacceptable toxicity
11. Life expectancy of at least 12 weeks.
12. WHO (ECOG) performance status <= 2, <= 1 if age > 75 years.
13. Adequate hepatic function
14. Adequate renal function

Exclusion Criteria:

1. Prior treatment with small molecule EGFR, HER2 or VEGFR tyrosine kinase inhibitors
2. Treatment with standard chemotherapy or cetuximab within the last 14 days
3. Treatment with bevacizumab within the last 28 days
4. History of other malignancies in the last 5 years, which could affect compliance with the protocol or interpretation of results. Patients with adequately treated basal or squamous cell skin cancer are generally eligible.
5. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality
6. Significant cardiovascular diseases
7. History of haemorrhagic or thrombotic event in the past 12 months. Known inherited predisposition to bleeds or to thrombosis.
8. Patient with history or clinical or radiological evidence of CNS disease or brain metastases.
9. Pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2007-11-01 (Actual)

PRIMARY OUTCOMES:
The RECIST criterion will be used to assess: objective response rate (PR + CR), and disease progression within the first 16 weeks | every 4 weeks
PFS | 16 weeks

SECONDARY OUTCOMES:
Progression-free survival (based on the RECIST criteria) | 66 Weeks
Overall survival | 66 Weeks
The incidence and intensity of Adverse Events with grading of Adverse Events according to the US NCI Common Terminology Criteria for Adverse Events (CTCAE version 3.0) | 66 Weeks
Changes in safety laboratory parameters | 66 Weeks
Effectiveness of dose reduction guidelines in managing adverse events | 66 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- France (24):
  - 1239.2.3305A clinique Saint Jean, Lyon
  - 1239.2.3305B Cabinet Médical, Lyon
  - 1239.2.3301A Hôpital Saint Antoine, Paris
  - 1239.2.3301B Hôpital Saint Antoine, Paris
  - 1239.2.3301C Hôpital Saint Antoine, Paris
  - 1239.2.3301D Hôpital Saint Antoine, Paris
  - 1239.2.3301E Hôpital Saint Antoine, Paris
  - 1239.2.3301F Hôpital Saint Antoine, Paris
  - 1239.2.3301G Hôpital Saint Antoine, Paris
  - 1239.2.3301H Hôpital Saint Antoine, Paris
  - 1239.2.3301I Hôpital Saint Antoine, Paris
  - 1239.2.3301J Hôpital Saint Antoine, Paris
  - 1239.2.3301K Hôpital Saint Antoine, Paris
  - 1239.2.3302A Hôpital Tenon, Paris
  - 1239.2.3302B Hôpital Tenon, Paris
  - 1239.2.3304A Hôpital Robert Debré, Reims
  - 1239.2.3304B Hôpital Robert Debré, Reims
  - 1239.2.3304C Hôpital Robert Debré, Reims
  - 1239.2.3303A Institut Gustave Roussy, Villejuif
  - 1239.2.3303B Institut Gustave Roussy, Villejuif
  - 1239.2.3303C Institut Gustave Roussy, Villejuif
  - 1239.2.3303D Institut Gustave Roussy, Villejuif
  - 1239.2.3303E Institut Gustave Roussy, Villejuif
  - 1239.2.3303F Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21737652